CLINICAL TRIAL: NCT05779163
Title: A Multicenter, Open Phase I/II Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of LBL-033 in the Treatment of Patients With Advanced Malignant Tumors.
Brief Title: A Phase I/II Clinical Trial of LBL-033 in the Treatment of Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanjing Leads Biolabs Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBL-033-CN001
Record Dates: First submitted 2023-03-07; First posted 2023-03-22 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Advanced Malignant Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LBL-033 (Experimental): LBL-033 for Injection; Initial dose - MTD; Q2W
  Interventions: Drug: LBL-033 for Injection

INTERVENTIONS:
Drug: LBL-033 for Injection — Initial dose - MTD; Q2W; intravenous infusion
  Other Names: LBL-033

SUMMARY:
This trial is an open and multicenter phase I/II clinical study, which aims to evaluate the safety, tolerability, PK characteristics, immunogenicity, and effectiveness.

DETAILED DESCRIPTION:
This is an open, multicenter Phase I/II clinical trial of LBL-033 in the treatment of patients with advanced malignant tumors，which aims to evaluate the safety, tolerability, PK characteristics, immunogenicity, and effectiveness.

The trial is divided into 2 parts: Phase 1 and Phase 2

Phase I study:

Dose-escalation and PK expansion.The PK expansion study will be judged on the basis of dose escalation data.

Phase II study:

Dose expansion included 4 cohorts that required patients with MUC16-positive malignancies.Blood samples will be collected from all subjects in this trial.

Phase I and Phase II studies are expected to recruit 113-468 patients

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the experimental treatment plan and visit plan, join the group voluntarily, and sign a written informed consent form;
2. Age ≥ 18 years old when signing the informed consent form;
3. The Eastern Cooperative Oncology Group's physical status scoring standard (ECOG) is 0~1;
4. The expected survival time is at least 12 weeks;
5. According to the evaluation of RECIST 1.1 standard, the subjects enrolled have at least one measurable Target lesion;
6. Subject has adequate organ and bone marrow function，Conforming to laboratory test results:
7. Males with fertility and females of childbearing age are willing to take effective contraceptive measures From the signing of the informed consent form to within 6 months after the last administration of the trial drug (including abstinence, intrauterine device, various hormonal contraception, correct use of contraception Sets，etc）; Women of childbearing age include pre-menopausal women and women within 2 years after menopause. Women of childbearing age must have a negative pregnancy test within 7 days before the first trial drug is administered.

Exclusion Criteria:

1. Have received other unmarketed clinical research drugs or treatments within 4 weeks before using the research drug for the first time;
2. Patients with active infection and currently requiring intravenous anti-infective treatment；
3. Those who have clinically uncontrollable pleural effusion, pericardial effusion , requiring repeated drainage or medical intervention;
4. The patient has a Medical history of immunodeficiency, including HIV antibody positive；
5. Women during pregnancy or lactation;
6. The investigator believes that the subject has other conditions that may affect compliance or are not suitable for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities（DLT） | At the end of Cycle 1（28 days after the first prespecified dose）
  DLT describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.
Maximum tolerated dose (MTD) | At the end of Cycle 1（28 days after the first prespecified dose）
  MTD is defined as the hightest dose level at which no more than 1 out of 6 subjects experiences a DLT during the first cycles

SECONDARY OUTCOMES:
Cmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy
  Maximum serum concentration
Tmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy
  After taking a single dose, Time to reach maximum plasma concentration
immunogenicity | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy
  The immunogenicity is evaluated by the incidence of anti-drug antibodies (ADA) and neutralizing antibodies (if applicable) in subjects
Disease Control Rate(DCR） | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy
  Percentage of participants achieving CR and PR and stable disease (SD).
Duration of Response(DOR） | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy
  The period from the participants first achieving CR or PR to disease progression.
Objective Response Rate (ORR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30 days after drug withdrawal or before the start of new anti-tumor therapy.
  Objective Response Rate (complete response (CR) + partial response (PR)), as assessed by Response Evaluation Criteria in Solid Tumors (RECIST 1.1), refers to the percentage of study subjects who achieve a complete response or partial response. This Secondary Outcome Measure was used for efficacy observations in Phase I study

CONTACTS AND LOCATIONS:
Overall Officials: jihong liu, Principal Investigator — Sun Yat-sen University
Locations (6):
- China (6):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - West China Second University Hospital,Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No